CLINICAL TRIAL: NCT01826604
Title: The Effect of a Barrier Self-Retaining Retractor in Obese Patients Undergoing Cesarean Section
Brief Title: Self-Retaining Retractor in Obese Patients Undergoing Cesarean Section
Acronym: Alexis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Katherine Scolari Childress, M.D., Principal Investigator, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22591
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Pregnancy; Obese
Keywords: cesarean section; Pregnant
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alexis O C-section retractor (Experimental): Alexis O C-section retractor will be used.
  Interventions: Device: Alexis O C-Section Retractor
- Control- Conventional retractors (Other): Conventional retractors for C-sections will be used.
  Interventions: Other: Control- Conventional retractors

INTERVENTIONS:
Device: Alexis O C-Section Retractor — The Alexis O C-section retractor will be used.
  Other Names: C-section dual ring retractor; Self retaining barrier retractor
  Arms: Alexis O C-section retractor
Other: Control- Conventional retractors — Conventional hand-held retractors will be used. A self-retaining barrier retractor will not be used.
  Other Names: Doyen retractor; Bladder blade; Richardson retractor
  Arms: Control- Conventional retractors

SUMMARY:
The purpose of this study is to investigate the effects of the Alexis O C-section retractor in obese patients (BMI ≥30 kg/m2) who undergo Cesarean sections. Patients will be randomized to the use of the Alexis retractor during Cesarean section (treatment group) or the use of traditional hand-held retractors (control group). We will determine if there is any difference in surgical site infection or wound disruption rates. We will also determine if there is a difference in the duration of surgery or length of time from skin incision to delivery of the infant, change in hemoglobin, estimated blood loss, and postoperative length of stay, intra-operative or postoperative anti-emetic requirements, need for hospital readmission or emergency room visits, or other complication rate between the two groups.

DETAILED DESCRIPTION:
This study will be a prospective randomized-controlled trial. It will take place at a single site at St. Mary's Health Center in Richmond Heights, Missouri. Pregnant women with a BMI ≥ 30 kg/m2 who will be undergoing non-emergent Cesarean sections for delivery will be eligible. Exclusion criteria will be patients who are undergoing emergency Cesarean section, patients who are in an immunosuppressed state (ie, HIV, cancer), if they have a pre-existing infection other than chorioamnionitis at the time of the Cesarean section, or have received steroids for more than two days. Chorioamnionitis will be defined by the presence of fever, uterine fundal tenderness, maternal tachycardia (>100 beats per minute), fetal tachycardia (>160 beats per minute), or purulent or foul-smelling vaginal discharge or amniotic fluid [15]. All Cesarean sections will be performed for standard indications and not for the purpose of the study. After informed consent is obtained in patients who choose to participate, patients will be randomly assigned to either the control group (conventional hand-held retractors used only) or to the treatment group (Alexis O C-section self-retaining retractor used as well as any hand held retractors that are deemed necessary by the surgeon). Both types of retractors are commonly used for cesarean sections in obese patients and the choice of retractor is made by physician preference. There will be no other differences between the two groups. Randomization will occur using a computer-generated randomization process prior to the start of the study and the individual assignments will be placed in opaque sealed envelopes. After a patient agrees to participate in the study, an envelope will be selected and opened to assign the patient to either the treatment or control group.

The Cesarean section will be performed for standard indications using standard surgical practice. All patients will receive pre-operative antibiotics according to St. Mary's Health Center standard practice. If the subcutaneous fat layer is >2 cm, it will be closed with a suture layer as is accepted standard practice. Both of these measures have been showed to be associated with decreased risk of postoperative surgical site infection and are standard practice [4, 16]. The depth of the subcutaneous fat layer will be measured during the surgery using the sterile ruler that is provided as part of the standard Cesarean section surgical instrument tray set. If the patient is assigned to the Alexis retractor group, the Alexis retractor will be placed once the peritoneal incision has been made and extended adequately. The peritoneal incision is part of the usual surgical technique during Cesarean sections. The Alexis retractor will then be placed with the outer ring positioned external to the incision overlying the skin, the internal ring positioned inside the peritoneum against the anterior abdominal wall, with the connecting clear plastic barrier retracting the abdominal wall. The abdominal cavity will be palpated to ensure no abdominal organs have been inadvertently incorporated into the retractor as is the accepted protocol when using the Alexis retractor. All other aspects of the Cesarean section will be done routinely. Patients will be blinded to whether they were in the control or the treatment group. Postoperative care will be the same for both groups, according to standard practice. Patients will be followed until 30 days postpartum. They will be instructed to follow up for a postoperative incision check 1-2 weeks postoperatively. Patients will be contacted by telephone 30 days postoperatively to inquire if they have developed any type of surgical site infection in the 30 days postoperatively. They will be informed of this process during the consent process. Surgical site infections will be defined using the CDC criteria [17]. Information will be collected from the patient's hospital and clinic chart, including patient demographic information (patient BMI, maternal age, race, gestational age at delivery, number of previous surgeries, gravidity, parity, and maternal comorbidities); neonatal outcomes (infant weight, APGAR scores, need for NICU admission); indication for cesarean section; if the patient was laboring; the presence or absence of ruptured membranes (and length of time if ruptured membranes present); positive or negative GBS culture; the presence of chorioamnionitis; type of skin and uterine surgery; total duration of surgery and duration from skin incision until delivery of the infant; occurrance and type of infection; number of days postoperatively an infection occurred; depth of subcutaneous fat layer, estimated blood loss during surgery; change in hemoglobin from admission to postoperative Day #1 (a lab for hemoglobin and hematocrit drawn on postoperative Day #1 after a Cesarean section is part of routine care); requirement of intra-operative and postoperative anti-emetics; type of skin closure performed; length of postoperative hospital stay; presence of postoperative infection or wound disruption during hospital admission; the need for postoperative antibiotics; and other postoperative complications. Information will also be collected from the one to two week postoperative check, including presence of infection or wound disruption, need for postoperative antibiotics, need for wound opening or exploration, visits to the Emergency Room or need for hospital readmission. Information will be collected during the postoperative telephone call that occurs 30 days after the procedure. Participants will be asked the same questions which is on the attached question sheet, and includes whether the patient experienced a diagnosis of a postoperative infection, need for postoperative antibiotics, visit to the Emergency Room or hospital readmission, or other complication within 30 days after the Cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* BMI greater than or equal to 30 kg/m squared
* Aged 14-50 years old
* Undergoing non-emergent cesarean section for delivery

Exclusion Criteria:

* Subjects undergoing emergency Cesarean-section
* Pre-existing concurrent infection other than chorioamnionitis
* State of immunosuppression (ie. HIV, cancer)
* Long-term steroid use (>2 days)
* Subjects with a BMI <30 kg/m2

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 301 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Scolari Childress, M.D., Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized controlled trial of obese women (BMI ≥30 kg/m2) undergoing non-emergent Cesarean section at St. Mary's Health Center, March 2013 to September 2014. Patients were randomized to the treatment group (using the Alexis O C-section retractor) or to the control group (using conventional hand-held retractors).
Pre-assignment Details: Non-emergent Cesarean delivery was defined by our institution's Cesarean section acuity scale, included those in which there was no immediate threat to the life of the patient or fetus. Not all Cesarean deliveries were elective, patients were included if there was typical time for routine Cesarean section preparation.
Groups:
- Alexis O C-section Retractor: The Alexis O C-section retractor will be used. Other hand-held retractors will be used as deemed necessary by the surgeon.
  Alexis O C-Section Retractor: The Alexis O C-section retractor will be used. Other hand-held retractors that are deemed necessary to the surgery by the physician will also be used.
- Control: Conventional hand-held surgical retractors used for C-sections will be used, including the bladder blade (Doyen retractor) and the Richardson retractor.
  Control- Conventional hand-held retractors: Conventional hand-held retractors will be used. A self-retaining barrier retractor will not be used.
Period: Overall Study
Arm/Group | Alexis O C-section Retractor | Control
Started | 144 | 157
Completed | 136 | 148
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Alexis O C-section Retractor: Alexis O retractor used during C-section
- Control: Other retractor used during C-section
- Total: Total of all reporting groups
Arm/Group | Alexis O C-section Retractor | Control | Total
Number analyzed (Participants) | 144 | 157 | 301
Age, Categorical [Count of Participants; unit: Participants] — Age of participants
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 144 | 157 | 301
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 28.5 [24.0 to 33.0] | 29 [24.5 to 32.0] | 28.8 [24.0 to 33.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 157 | 301
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 144 | 157 | 301
Gravidity [Mean (Full Range); unit: live births] | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
BMI [Median (Full Range); unit: kg/m2] — BMI mean
  kg/m2 | 39.9 [35.6 to 45.6] | 40.6 [34.9 to 46.5] | 40.1 [34.9 to 46.5]
Subcutaneous thickness [Median (Full Range); unit: cm] | 3.0 [2.0 to 4.0] | 3.0 [2.3 to 4.0] | 3.0 [2.0 to 4.0]
Chorioamnionitis [Number; unit: participants] — Not all participants had chorioamnionitis-this accounts for the difference from baseline numbers
  participants | 8 | 6 | 14
Group beta streptococcus colonization [Number; unit: participants] — Not all participants were positive for GBS-this accounts for the difference from baseline numbers
  participants | 38 | 49 | 87
Low transverse-skin incision [Number; unit: participants] — Not all participants had a low transverse skin incision-this accounts for the difference from baseline numbers
  participants | 130 | 144 | 274
Low transverse-Uterine incision [Number; unit: participants] — Not all participants had a low transverse uterine incision-this accounts for the difference from baseline numbers
  participants | 135 | 144 | 279
Tobacco Use [Number; unit: participants] | 27 | 46 | 73

OUTCOME MEASURES:

1. Primary Outcome: Wound Infection or Disruption
Description: We will compare the number of patients with wound infections or disruptions when the Alexis O C-Section retractor is used vs when it is not used.
Time Frame: Time of surgery to 30 days post op
Population: Any SSI or wound disruption during 30 day postoperative period
Measure: Number; unit: participants
Groups:
- Alexis Retractor; Control: Outcomes at each time period are additive so that patients who experienced the outcome at each time point are included in the next time point. Patients may have experienced more than one type of outcome and are reported for each outcome experienced. The outcome of SSI or wound disruption includes cumulative of all patients who experienced either type of outcome.
Arm/Group | Alexis Retractor | Control
Number analyzed (Participants) | 136 | 148
participants | 38 | 37

2. Secondary Outcome: Secondary Outcomes Will Include the Differences Between the Two Groups.
Description: Secondary outcomes will include the duration of surgery or length of time from skin incision to delivery of the infant, change in hemoglobin, estimated blood loss, and postoperative length of stay, intra-operative or postoperative anti-emetic requirements, need for hospital readmission or emergency room visits, or other complication rates between the two groups.
Time Frame: From the time of surgery to 30 days post-op.
Population: infection during 30 day postoperative period
Measure: Number; unit: participants
Arm/Group | Alexis Retractor | Control
Number analyzed (Participants) | 28 | 26
participants
  Surgical site infection during 30 day postop | 20 | 19
  Superficial incisional during 30 day postop | 14 | 13
  Deep organ/space during 30 day postop | 6 | 6
  Wound disruption during 30 day postop | 18 | 18

ADVERSE EVENTS:
Time Frame: 6 months post op
Groups:
- Alexis Retractor; Control: No adverse events
Arm/Group | Alexis Retractor | Control
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/157
Other Adverse Events (participants affected / at risk) | 0/144 | 0/157

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes